CLINICAL TRIAL: NCT01090206
Title: Correlation Between Vitamin D Status and Bone Mineral Density in Patients With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PT 104212
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Hemophilia A; Hemophilia B; Vitamin D Deficiency
Keywords: Hemophilia; Vitamin D
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Vitamin D Deficiency | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemophilia, Vitamin D deficiency (Other): 1. Hemophilia, Rickets - Vitamin D per endocrine consult
  2. Hemophilia, Vitamin D deficient - Vitamin D 2000 units daily plus calcium
  3. Hemophilia, Normal Vitamin D - no intervention - observation only
  Interventions: Dietary Supplement: Vitamin D and calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D and calcium — Doses will be based on Vitamin D levels

SUMMARY:
Study will look at baseline Vitamin D levels, calcium, albumin, liver enzymes, testosterone, osteocalcin, urine N telopeptides, bone mineral density, nutritional assessment and physical activity assessment of boys with hemophilia A or B (ages 2-20 yrs). Patients with low vitamin D levels will receive therapeutic doses of Vitamin D. At end of one year follow up studies will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Hemophilia A or B
* ages 2-21 years

Exclusion Criteria:

* therapeutic vitamin D or calcium supplementation within 3 months of study entry

Ages: 2 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Correlate between Vitamin D deficiency, low bone mass and lack of weight bearing physical activity | 1year

SECONDARY OUTCOMES:
Determine bone mass (density) in hemophilia patients | 1 yr
establish dose and duration of treatment with vitamin D | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Gita V Massey, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States